CLINICAL TRIAL: NCT02564367
Title: Multicenter Phase I/II Feasibility Study of Adjuvant Treatment With S-1 in Patients After R0-Resection of Adenocarcinoma of the Stomach and Esophagogastric Junction
Brief Title: Feasibility Study of Adjuvant Treatment With S-1 in Patients After R0-Resection of Adenocarcinoma of the Stomach and Esophagogastric Junction
Acronym: S-1 adjuvant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Nordic Pharma SAS (Industry); Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMBH-STO-0114; 2014-004116-11 (EudraCT Number)
Record Dates: First submitted 2015-04-10; First posted 2015-09-30 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Adenocarcinoma,Stomach; Adenocarcinoma, Esophagogastric Junction
MeSH Terms: conditions — Adenocarcinoma | interventions — S 1 (combination); tegafur-gimeracil-oteracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): First Cohort 1:
  (n = 30 patients) 18 cycles S-1
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — 18 cycles S-1, orally administered twice daily D1-14, q 3 wks
  S-1 starting dose: 2 x 30 mg/m^2 body surface area (BSA), D1-14, q 3 wks First dose reduction: 2 x 25 mg/m^2 BSA, D1-14, q 3 wks Second dose reduction: 2 x 20 mg/m^2 BSA, D1-14, q 3 wks
  Other Names: Teysuno

SUMMARY:
Multicenter trial in Germany:

Feasibility Study of Adjuvant Treatment with S-1 in Patients after R0-Resection of Adenocarcinoma of the Stomach and Esophagogastric Junction with the aim to show the feasibility and tolerability of adjuvant S-1 treatment in Caucasian patients and to determine the recommended dose for the treatment regimen.

DETAILED DESCRIPTION:
Patients will be enrolled in one cohorts.

Cohort 1 consists of 30 patients who receive S-1 twice daily for 18 cycles (D1-14 q 3 wks).

ELIGIBILITY:
Inclusion Criteria:

1. Patient signed and dated informed consent before the start of any specific protocol procedures
2. Adult Caucasian patients ≥ 18 years of age
3. Histologically confirmed diagnosis of adenocarcinoma of the stomach and esophagogastric (EG) junction classified as uT2/uT3/uT4, any N category, M0 or any uT, N+, M0 patient (for patients having received neoadjuvant chemotherapy) or pT2/pT3/pT4, any N category, M0 or any pT, N+, M0 (for patients having received primary surgery) according to Union international contre le cancer (UICC) TNM edition 7.
4. R0-resection after neoadjuvant treatment. However, patients can also be included if neoadjuvant treatment could not be performed due to medical indication of primary surgery (perforation, bleeding etc.) or was not performed due to understaging.
5. D2 lymph node dissection performed
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
7. Consent to translational research being performed on tumor tissue of the primary tumor that had been removed during the resection surgery. Translational research will be performed only upon completion of routine histological and pathological evaluations of the tumor
8. Females of childbearing potential (FCBP) must have a negative pregnancy test within 7 days of the first application of study treatment and must agree to use effective contraceptive birth control measures (Pearl Index < 1) during the course of the trial and for at least 6 months after last application of S-1.

   Females of childbearing potential (FCBPs) should be included after a confirmed menstrual period (only if applicable, i.e. still having menses) and must have a negative highly sensitive pregnancy test within 7 days prior to the first application of study treatment and must agree to use highly effective contraceptive birth control measures (Pearl Index < 1) during the course of the trial and for at least 6 months after last application of S-1.

   Such highly effective birth control methods include:
   * oral, intravaginal, or transdermal combined hormonal contraception associated with inhibition of ovulation
   * oral, injectable, or implantable progesterone-only hormonal contraception associated with inhibition of ovulation
   * intrauterine device
   * intrauterine hormone-releasing system
   * bilateral tubal occlusion
   * commitment to complete abstinence from heterosexual contact

   A female subject following menarche is considered to be of childbearing potential unless she is naturally amenorrhoeic for ≥ 1 year without an alternative medical reason, or unless she is permanently sterile (permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy).
9. Males must agree not to father a child during the course of the trial and for at least 6 months after last administration of S-1 and must agree to use condoms during the course of the trial and for at least 6 months after last administration of S-1 in case of sexual intercourse with FCBP or pregnant female.
10. Patient must be able to take medication orally within eight weeks after surgery at the start of S-1.
11. Normal cardiac function demonstrated by Electrocardiogram (ECG) and echocardiogram (LVEF ≥ 55%)
12. Adequate bone marrow, hepatic and renal function defined as

    * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L
    * Haemoglobin ≥ 9 g/dL
    * Platelets ≥ 100 x 10^9/L
    * Albumin ≥ 2.5 g/dL
    * Total bilirubin ≤ 2 mg/dL
    * GOT/AST and GPT/ALT ≤ 3 x Upper normal limit (ULN)
    * Calculated creatinine clearance according to MDRD equation ≥ 50 mL/min
13. Patient's legal capacity to consent to study participation

Exclusion Criteria:

1. Metastatic disease (exclusion of metastatic disease by a postoperative CT or MRI scan of thorax and abdomen within 3 weeks prior to start of adjuvant therapy)
2. Polyneuropathy > grade 1 (NCI CTCAE version 4.0)
3. Evidence of ascites or liver cirrhosis
4. Patient is pregnant or breast-feeding
5. Patient underwent a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment, or there is an anticipated need for major surgical procedure during the course of the study.
6. Heart failure ≥ NYHA functional classification system grade 2
7. Myocardial infarction, unstable angina, cardiac angioplasty or stenting procedure within the last 6 months.
8. Medical history of pulmonary fibrosis or interstitial lung disease (ILD)
9. Active or uncontrolled bacterial, viral, or fungal infection that requires systemic treatment
10. Known HIV-, HBV-, and HCV-infection
11. Concurrent disease or condition that would make the patient inappropriate for study participation or would interfere with the patient's safety.
12. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
13. Any cancer therapy (chemotherapy, radiation therapy, biologic therapy, immunotherapy, or hormonal therapy) after resection surgery or requirement for concurrent cancer treatment during study treatment with S-1.
14. Participation in another clinical trial or treatment with an investigational drug after surgery and during study treatment with S-1.
15. Known immediate or delayed hypersensitivity to any of the active substances of S-1 (tegafur, gimeracil, and oteracil) or to any of the excipients or to drugs chemically related to S-1 (e.g. 5-fluorouracil)
16. History of severe and unexpected reactions to fluoropyrimidine therapy
17. Known dihydropyrimidine dehydrogenase (DPD) deficiency
18. Treatment with DPD inhibitors, including sorivudine or its chemically related analogues such as brivudine within 4 weeks before start of study drug or during study treatment
19. Previous or concurrent malignant tumor disease other than underlying tumor disease with the exception of cervical cancer in situ, adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, superficial bladder tumors (Ta, Tis, and T1) or any curatively treated tumors > 5 years prior to enrolment
20. Known alcohol abuse or drug addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
number of patients with discontinuation of S-1 due to intolerable adverse reactions | 12 months

SECONDARY OUTCOMES:
One-year relapse-free survival rate | 12 months
  Mo local relapse or distant metastases within one year after start of adjuvant treatment
Relapse-free survival | 2 years
  relapse-free survival until end of study
Quality of life | 12 months
  European Organisation for Research and Treatment of Cancer (EORTC) C30 questionnaires
One-year survival rate | 1 years
Overall survival | 2 years

OTHER OUTCOMES:
plasma concentration of Tegafur (FT) | 12 months
  To evaluate the pharmacokinetics of FT
plasma concentration of 5-Fluorouracil (5-FU) | 12 months
  To evaluate the pharmacokinetics of 5-FU
plasma concentration of Gimeracil (CDHP) | 12 months
  To evaluate the pharmacokinetics of CDHP

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, Prof. Dr., Principal Investigator — Klinikum der Universität München, Campus Großhadern
Locations (1):
- Klinikum der Universität München, Campus Großhadern, München, Bavaria, Germany